CLINICAL TRIAL: NCT02423629
Title: Agili-C™ Implant Performance Evaluation in the Repair of Cartilage and Osteochondral Defects (OCD)
Brief Title: Agili-C™ Implant Performance Evaluation in the Repair of Cartilage and Osteochondral Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0019
Record Dates: First submitted 2014-12-03; First posted 2015-04-22 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2019-10

CONDITIONS: Cartilage or Osteochondral Defects in the Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Agili C™ (Other): Candidates will be screened for possible inclusion in the trial. Candidates that are approved by the adjudication committee will be considered for study enrollment and then operated. Note: in case intra-operatively a medical condition is observed which is not aligned with the inclusion/exclusion criteria, the Subject will not be implanted with the Agili-C™ device and will not be considered enrolled in the study.
  Interventions: Device: Agili-C™ implantation procedure

INTERVENTIONS:
Device: Agili-C™ implantation procedure — Candidates for Agili-C™ implantation will be screened for possible inclusion in the trial. Candidates that are approved by the adjudication committee will be considered for study enrollment and then operated. Note: in case intra-operatively a medical condition is observed which is not aligned with the inclusion/exclusion criteria, the Subject will not be implanted with the Agili-C™ device and will not be considered enrolled in the study.

SUMMARY:
Evaluate the performance of the Agili-C™ in the repair of Cartilage and Osteochondral defects.

DETAILED DESCRIPTION:
Agili-C™ implant is a CE marked, bi-phasic, porous resorbable tissue regeneration scaffold for the treatment of articular cartilage and/or osteochondral defects.

The Agili-C™ implant will be implanted using the Agili-Kit™ surgical toolset which is designed for the precise preparation of sites in cartilage and osteochondral defects, for implanting the Agili-C™ implant

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Up to 3 treatable cartilage lesions, ICRS IIIa - IVb on the femoral condyles or the trochlea,
3. Symptomatic total treatable area 1-7 cm2. Asymptomatic lesions will not be included in the calculation
4. KOOS Pain score at baseline is not less than 30 and not more than 65
5. Must be physically and mentally willing and able to comply with post- operative rehabilitation protocol and scheduled clinical and radiographic visits.
6. Informed consent signing

Exclusion Criteria:

1. Bony defect depth deeper than 8mm, according to imaging Articular cartilage lesions in the tibia or the patella, ICRS grades IVa and IVb
2. Any previous ligamentous repair or malalignment correction in the index knee within the last 3 months
3. Significant instability of the index knee according to IKDC Knee Examination Form 2000, Grade C (abnormal) or D (severely abnormal)
4. Lack of functional remaining meniscus
5. Meniscal transplantation in the past 6 months
6. Malalignment more than 5 degrees varus OR 5 degrees valgus according to standing X-ray
7. Any known tumor of the index knee
8. Any know history of infection of the index knee
9. Any known history of inflammatory arthropathy or crystal-deposition arthropathy
10. Any known systemic cartilage and/or bone disorder such as but not limited to chondrodysplasia or osteogenesis imperfecta
11. Body mass index >35
12. Osteoarthritis of the index knee graded as 4 according to the Kellgren- Lawrence scale
13. Chemotherapy treatment in the past 12 months
14. Any previous surgical cartilage treatment in the index knee within the last 6 months
15. History of allergic reaction or intolerance of materials containing calcium carbonate or hyaluronate
16. Patient who is pregnant or intends to become pregnant during the study
17. History of any significant systemic disease, such as but not limited to, HIV infection, hepatitis infection or HTLV infection; known coagulopathies, that might compromise the subject's welfare
18. Known substance abuse or alcohol abuse
19. Participation in other clinical trials within 30 days prior to the study or concurrent with the study
20. Known insulin dependent diabetes mellitus
21. Unable to undergo MRI or X-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-05; Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
• The KOOS Pain Subscale relative to baseline | 24 Months
  The KOOS pain subscale is evaluated at 6m, 12m, 18m & 24m

SECONDARY OUTCOMES:
• Improvement in other KOOS subscales relative to baseline | 24 Months
  Other KOOS subscales are evaluated at 6m, 12m, 18m & 24m
• Improvement in IKDC Subjective Knee Score relative to baseline | 24 Months
  IKDC Subjective Knee Score is evaluated at 6m, 12m, 18m & 24m
• Improvement in SF-36 Survey | 24 Months
  SF-36 Survey is evaluated at 6m, 12m, 18m & 24m
• Improvement in Tegner Score | 24 Months
  Tegner Score is evaluated at 6m, 12m, 18m & 24m
• Improvement in Lysholm Knee Scoring Scale | 24 Months
  Lysholm Knee Scoring Scale is evaluated at 6m, 12m, 18m & 24m
• Joint Space maintenance rate according to X-ray | 24 Months
  Joint Space maintenance rate is evaluated at 12m & 24m
• Defect Fill according to MRI | 24 Months
  Defect Fill according to MRI is evaluated at 6m, 12m, 18m & 24m
Improvement of Overall KOOS (average of all KOOS Subscales) relative to baseline | 24 mMonths
  The KOOS Overall is evaluated at 6, 12,18 & 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — Rizzoli Institute, Bologna , Italy
Locations (8):
- Medical University of Vienna, Vienna, Austria
- AZ Monica, Antwerp, Belgium
- Hasharon medical center, Petah Tikva, Israel
- Rizzoli Orthopaedic Institute, Bologna, Italy
- Specialist Hospital. Louis Rydygier, Krakow, Poland
- Timişoara County Hospital, Timișoara, Romania
- Institut za Ortopedsko-hirurške Bolesti "banjica", Belgrade, Serbia
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No